CLINICAL TRIAL: NCT03855397
Title: Pain and Safety of Microneedle Application in the Oral Cavity of Human Volunteers
Brief Title: Pain and Safety of Microneedles in Oral Cavity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Principal Investigator, Michelle Franz Montan Braga Leite, DDS, MSc, PhD, Principal Investigator, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAAE: 42926115.3.0000.5418
Record Dates: First submitted 2019-01-29; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-01

CONDITIONS: Oral Cavity Disease
Keywords: Microneedles; Buccal mucosa; Transbuccal administration
MeSH Terms: conditions — Mouth Diseases | interventions — PittCoVacc; Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microneedles (Experimental): Application of microneedle patch, 30G hypodermic needle (positive control) and flat patch (negative control) in the lip, buccal, tongue, palatal and gingival mucosa for pain and safety assessment
  Interventions: Other: Microneedle; Other: Hypodermic needle; Other: Flat patch

INTERVENTIONS:
Other: Microneedle — A microneedle patch (no drug) was applied in the following oral cavity sites: lip, buccal, tongue, palatal and gingival mucosa to access pain, discomfort and safety.
Other: Hypodermic needle — 30 gauge hypodermic needle was inserted in the following oral cavity sites: lip, buccal, tongue, palatal and gingival mucosa.
  Other Names: positive control
Other: Flat patch — A flat patch was applied in the following oral cavity sites: lip, buccal, tongue, palatal and gingival mucosa.
  Other Names: negative control

SUMMARY:
A randomized, crossover, double-blind, placebo-controlled, one-session clinical trial with 30 male volunteers was performed to access pain and safety of microneedle topical application in different regions of the oral cavity.

DETAILED DESCRIPTION:
A randomized, crossover, double-blind, placebo-controlled, one-session clinical trial with 30 male volunteers was performed by applying a microneedle patch in the following regions of the oral cavity: lip (inner lower), buccal (cheek: 1 cm behind the month angle), tongue (dorsal surface), hard palate (anterior region), and attached gingiva (between central and lateral upper incisors). A 30 gauge hypodermic needle and an identical patch but without microneedles sticking out, were used as positive and negative controls, respectively. The application force was standardized to 10N by an applicator composed of a 5 mL syringe and a spring. Insertions were performed with a gap of 30 seconds. Pain and discomfort associated to the procedure was evaluated with a Visual Analogue Scale (VAS), by a blinded-dentist. The safety associated to microneedle application was verified immediately after the application (0h) and after the next day (24h). The different application sites were inspected visually for bleeding, ulceration, bruising, redness or swelling.

ELIGIBILITY:
Inclusion Criteria:

- Healthy male

Exclusion Criteria:

- Volunteers were free from cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal and haematological diseases, psychiatric disorders, smokers or alcoholic.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-12-16 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity assessment by Visual Analogue Scale after microneedle application in the oral cavity | 30 seconds
  Pain was evaluated after microneedles, hypodermic needle or negative control topical application application in different oral cavity sites
Number of participants with treatment-related adverse events as assessed by visual inspection of ecchymosis, ulceration, redness, swelling or bleeding after microneedles use in the oral cavity | 24 hours
  Any sign of ecchymosis, ulceration, redness, swelling or bleeding right after and 24 h later applications of the devices in different oral cavity sites

SECONDARY OUTCOMES:
Confirmation of mucosal perforationin the oral cavity after application of the devices | Right after microneedle application
  Mucosal perforation after microneedles application was confirmed by applying gentian violet to stain the sites of microneedle insertion

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Leite, PhD, Principal Investigator — University of Campinas, Brazil; Harvinder S Gill, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Michelle Franz Montan Braga Leite, Piracicaba, São Paulo, Brazil